CLINICAL TRIAL: NCT07379970
Title: Effects of Wearable Device Functions and Health Coaching on Device-measured Movement Behaviours and Cardiometabolic Risk Factors in Adults With Central Obesity: a Randomised Controlled Trial
Brief Title: Effects of Wearable Device Functions and Health Coaching on Device-measured Movement Behaviours and Cardiometabolic Risk Factors in Adults With Central Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Kim, Youngwon, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: healthcoachingrct
Record Dates: First submitted 2026-01-15; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Fitness Trackers; Cardio Vascular Disease; Physical Activities; Exercise; Health Coaching
Keywords: movement behavior; NDPP Program; randomized controlled trial; wearable technology
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: parallel-group, open randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Group allocation will be concealed from study staff until the 7-day pre-intervention period begins (for preparation of corresponding e-leaflets, lifestyle coaching courses and baseline Fitbit step goal calculations), and from participants until the interventions are delivered. Given the nature of the interventions delivered, it will be impossible for participants to be blinded to the specific intervention they receive once the initial interventions are provided; however, study staff analyzing participants' de-identified data will remain blinded to participant randomization assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care Control (No Intervention): Participants will continue their usual lifestyle without receiving a wearable device or behavioral intervention.
- Fitbit Only (Experimental): Participants will receive a Fitbit wearable device and use selected Fitbit functions related to physical activity and sleep.
  Interventions: Device: Fitbit Wearable Device
- Fitbit + Lifestyle Coaching (Experimental): Participants will receive a Fitbit wearable device and participate in a structured lifestyle coaching program adapted from the U.S. CDC National Diabetes Prevention Program (NDPP).
  Interventions: Behavioral: Lifestyle Coaching Program

INTERVENTIONS:
Device: Fitbit Wearable Device — Participants will use a Fitbit wearable device with the following evidence-based functions enabled: step goal setting (10% higher than baseline daily steps), sleep goal setting (8 hours per day), activity prompts (vibration alert when fewer than 250 steps are accumulated per hour), and community features such as activity or exercise challenges. These functions support self-monitoring, goal setting, prompts, feedback, and social support.
  Arms: Fitbit Only
Behavioral: Lifestyle Coaching Program — Participants will receive a structured lifestyle coaching program adapted from the U.S. Centers for Disease Control and Prevention National Diabetes Prevention Program (NDPP). The program includes at least 22 coaching sessions delivered over approximately 12 months. Sessions focus on cardiometabolic disease risk factors, goal setting, self-monitoring of physical activity, sleep, diet, and stress, strategies to initiate and maintain healthy behaviors, social support, and review of progress and challenges.
  Arms: Fitbit + Lifestyle Coaching

SUMMARY:
This study is a randomized controlled trial. The objective of this study is to investigate:

1. the effects of 1-year evidence-based interventions incorporating wearable device functions alone on device-measured movement behaviours and cardiometabolic risk factors among adults with central obesity; and
2. the effects of 1-year evidence-based interventions incorporating wearable device functions combined with health coaching on device-measured movement behaviours and cardiometabolic risk factors among adults with central obesity.

We hypothesise that the use of wearable device functions in combination with health coaching will lead to significantly greater improvements in device-measured movement behaviours and cardiometabolic risk factors compared with no intervention and wearable device functions alone, both after the 12-month intervention and at the 6-month follow-up.

This study will implement a parallel-group, open-label, 1-year randomized controlled trial involving 133 adults aged 40 years or older with central obesity. The trial will examine the effects of a cutting-edge intervention using evidence-based wearable device functions alone or in combination with evidence-based health coaching on movement behaviours and cardiometabolic risk factors.

All participants will provide written informed consent prior to participation and will be informed that they may withdraw from the study at any time during the study period. A staff member without access to participant information will generate a computer-based randomization list using permuted blocks of six, with two participants allocated to each of the three groups (two intervention groups and one control group) per block, in a 2:2:2 allocation ratio.

The control group will not receive a Fitbit device and will be asked to continue their usual lifestyle. The two intervention groups will use four evidence-based Fitbit functions: step goal setting, sleep goal setting, activity prompts, and community functions. The key difference between the two intervention groups is that one group will additionally receive a structured health coaching program adapted from the U.S. Centers for Disease Control and Prevention (CDC) National Diabetes Prevention Program (NDPP), as used in our prior trial.

The CDC NDPP recommends that at least 22 health coaching sessions be delivered over a 1-year period, depending on participants' needs, and provides corresponding curricula and handouts outlining session content. Coaching sessions will be delivered by trained research staff who have received appropriate professional training in health coaching delivery.

The lifestyle change program will include, but not be limited to:

1. education on cardiometabolic disease risk factors (e.g., type 2 diabetes, coronary heart disease, and stroke);
2. goal planning and goal setting;
3. strategies for self-monitoring physical activity, sleep, diet, and stress;
4. strategies for initiating and maintaining favourable levels of physical activity, diet, and sleep;
5. strategies for obtaining support from family, friends, and co-workers; and
6. review of achievements and challenges during the intervention period, with goal setting and planning for the subsequent 6-month follow-up period.

Participants will attend the research laboratory on three occasions: at baseline, immediately after the 12-month intervention, and at the 6-month follow-up. Assessments will include demographic information, standing height, body weight, body mass index, waist circumference, hip circumference, waist-to-hip ratio, systolic and diastolic blood pressure, and questionnaires.

At each laboratory visit, one EDTA blood sample and one clotted blood sample will be collected by a trained phlebotomist and analysed by an accredited medical diagnostic centre to assess cardiometabolic risk markers, including total cholesterol, HDL cholesterol, LDL cholesterol, and triglycerides.

An Axivity AX6 device will be used as a research-grade accelerometer to assess movement behaviours, including sleep, sedentary time, light physical activity, moderate-to-vigorous physical activity (MVPA), steps, energy expenditure, and resting heart rate. Participants will also be asked to wear the Axivity device on the dominant wrist for seven consecutive days at baseline and post-intervention.

Research staff will access participants' Fitbit web accounts to extract Fitbit data, activate Fitbit functions for the intervention groups, and monitor device battery life. Reminders to wear and charge the Fitbit and research-grade accelerometer will be sent every seven days via WhatsApp to promote protocol compliance. To further support adherence, participants who complete all study assessments will receive a HKD 500 supermarket voucher.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* Central obesity, defined as waist circumference: ≥90 cm for men; ≥80 cm for women
* Insufficient physical activity based on World Health Organization (WHO) guidelines
* Physical activity assessed using the International Physical Activity Questionnaire (IPAQ) - Short Form
* Ownership of a smartphone
* Able to read and understand English or Chinese

Exclusion Criteria:

* unable to perform daily-life activities, based on the Physical Activity Readiness-Questionnaire (PAR-Q) (24) and/or participation in another lifestyle-change intervention study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
24-hour Movement Behavior Composition (Accelerometer-derived) | Baseline, 12-month post-intervention
  The primary outcome is the 24-hour composition of movement behaviors, defined as the relative distribution of time spent in sedentary behavior, light physical activity, moderate-to-vigorous physical activity (MVPA), and sleep within a 24-hour period. These components will be derived from accelerometer data and jointly analyzed as a single compositional outcome using compositional data analysis methods.

SECONDARY OUTCOMES:
Body Weight | Baseline, 12 months
  Body weight measured using a calibrated digital scale. Unit of Measure: Kilograms (kg)
Waist Circumference | Baseline, 12 months
  Waist circumference measured at the midpoint between the lowest rib and the iliac crest. Unit of Measure: Centimeters (cm)
Blood Pressure | Baseline, 12 months
  Systolic and diastolic blood pressure measured using a standardized BP monitor. Unit of Measure: mmHg
Blood Lipid Profile | Baseline, 12 months
  Total cholesterol, HDL cholesterol, LDL cholesterol, and triglycerides measured from fasting blood samples. Unit of Measure: mmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Physiology Lab, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The datasets analysed during the current study and statistical code are available from the corresponding author on reasonable request, as is the full protocol.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The datasets analysed during the current study and statistical code will be available after the completion of the study
Access Criteria: IPD data can be accessed based on reasonable request by contacting the corresponding author.